CLINICAL TRIAL: NCT05524662
Title: Clinical and Histological Evaluation of BTL-785F Device for Non-invasive Treatment of Face
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BTL Industries Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BTL-785_CTUS900
Record Dates: First submitted 2022-08-30; First posted 2022-09-01 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Wrinkle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- BTL-785-7 Treatment (Experimental): Subjects will be enrolled for an active treatment with BTL-785F device (BTL-785-7 applicator) for non-invasive facial rejuvenation.
  Interventions: Device: BTL-785-7
- Control (No Intervention): One subject will serve as a control.

INTERVENTIONS:
Device: BTL-785-7 — Treatment with BTL-785F device (BTL-785-7 applicator) for non-invasive facial rejuvenation.
  Arms: BTL-785-7 Treatment

SUMMARY:
This study will evaluate the clinical efficacy, safety and the performance of the BTL-785-7 applicator of the BTL-785F system for non-invasive treatment of facial wrinkles and overall improvement of facial appearance.

DETAILED DESCRIPTION:
The changes in the skin related to the connective tissue structural proteins (i. e. elastin and collagen fibers) will be assessed histologically. The study is a prospective, single-center, two-arm, open-label study. The subjects will be enrolled and assigned into two groups; Group A (RF & EMF) and Control group, which will not receive any treatment.

At the baseline visit, health status will be assessed. Inclusion and exclusion criteria will be verified and informed consent will be signed. Punch biopsies of the facial skin (preauricular area) for the examination of changes related to skin's connective tissue, and photographs of the treated area will be taken.

The treatment administration phase in the treatment group will consist of four (4) treatment visits, delivered 5-10 days apart.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects over 21 years of age seeking treatment for reduction of wrinkles and overall aesthetic improvement of the face
* Subjects should be able understand the investigative nature of the treatment, the possible benefits and side effects, and must sign the Informed Consent Form
* Presence of clearly visible wrinkles in the treated area when the face is relaxed as deemed appropriate by the Investigator
* Subjects willing and able to abstain from partaking in any facial treatments other than the study procedure during study participation
* Willingness to comply with study instructions, to return to the clinic for the required visits, to undergo punch biopsies and to have photographs of their face taken

Exclusion Criteria:

* Bacterial or viral infection, acute inflammations ,
* Impaired immune system
* Isotretinoin in the past 12 months
* Skin related autoimmune diseases
* Radiation therapy and chemotherapy
* Poor healing and unhealed wounds in the treatment area
* Metal implants
* Permanent implant in the treated area
* Pacemaker or internal defibrillator, or any other active electrical implant anywhere in the body
* Facial dermabrasion, facial resurfacing, or deep chemical peeling in the treatment area within 3 months prior to the treatment
* Current or history of skin cancer, or current condition of any other type of cancer, or pre-malignant moles
* History of any type of cancer
* Active collagen diseases
* Cardiovascular diseases (such as vascular diseases, peripheral arterial disease, thrombophlebitis and thrombosis)1
* Pregnancy/nursing or IVF procedure
* History of bleeding coagulopathies, use of anticoagulants
* Any active condition in the treatment area, such as sores, psoriasis, eczema, rash and rosacea
* Any surgical procedure in the treatment area within the last three months or before complete healing
* Poorly controlled endocrine disorders, such as diabetes
* Electroanalgesia without exact diagnosis of pain etiology
* Serious psychopathological disorders (such as schizophrenia)
* Neurological disorders (such as multiple cerebrospinal sclerosis, epilepsy)
* Blood vessels and lymphatic vessels inflammation

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2022-12-10 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Histological examination | 5 months
  Evaluation of the facial skin to assess the changes related to connective tissue structural proteins in the biopsies obtained from the treatment group and control. Subjects will have one 3 mm punch biopsy obtained at the baseline and subsequent biopsies at the follow-up visits.

SECONDARY OUTCOMES:
Subject Satisfaction | 5 months
  The 7-point Likert scale Subject Satisfaction Questionnaire will be used for evaluating the satisfaction. The Subject Satisfaction Questionnaire will be given to subjects after the last therapy, at 1-month and 3-month follow-up. The answers to the questions related to the subjects' overall skin and face appearance will vary from "strongly agree" to "strongly disagree".
Therapy Comfort | 5 months
  The 7-point Likert scale Therapy Comfort questionnaire will be used for evaluating the comfort during the treatment sessions. Pain sensation will be rated by the subjects from 0 (no pain) to 10 (worst possible pain).
Evaluation of Wrinkle Severity | 5 months
  Three independent evaluators will evaluate changes of wrinkle severity according to the Fitzpatrick Wrinkle and Elastosis Scale (FWES) using the photographs of treated areas for wrinkles (left and right cheeks and the forehead) taken at the baseline, last therapy visit and each follow-up visit. Wrinkle severity improvement according to FWES is considered when there is a decrease in score of the scale. The baseline and post-treatment scores will be compared. If applicable, the statistical significance of obtained results will be analyzed in Microsoft Excel spreadsheet software. The level of significance (α) will be set as 5%.
Evaluation of Overall Facial Appearance According to GAIS | 5 months
  Three evaluators will evaluate facial appearance in the treatment group according to the Global Aesthetic Improvement Scale (GAIS) using the photographs taken at the baseline, last therapy visit and both follow-up visits. Each evaluator will be asked to assign a score to a set of photographs. Facial appearance improvement to GAIS is considered when there is an increase in score of the scale. The baseline and post-treatment scores will be compared. If applicable, the statistical significance of obtained results will be analyzed in Microsoft Excel spreadsheet software. The level of significance (α) will be set as 5%.

CONTACTS AND LOCATIONS:
Locations (1):
- Schweiger Dermatology PC, Reseach Division, Hackensack, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No